CLINICAL TRIAL: NCT06724341
Title: Effect of Active and Passive Augmented Reality Glasses in Behavioral Children Management for Inferior Alveolar Nerve Block - A Randomized Controlled Trial
Brief Title: Impact of AR Glasses on Children's Behavior During Dental Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Pedo-05-2024
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Anaesthesia; Anxiety
Keywords: Complementary Therapies; Pediatric Dentistry; Behavior Management; Augmented Reality Glasses
MeSH Terms: conditions — Anxiety Disorders | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group: inferior alveolar nerve block will be administrated with passive behavior management (Experimental)
  Interventions: Behavioral: Distraction
- Movies group: inferior alveolar nerve block will be administrated with displaying animated movies di (Experimental)
  Interventions: Behavioral: Distraction
- Video games group: Application of active behavior management by usage video games on the screen of a (Experimental)
  Interventions: Behavioral: Distraction
- Movies and Video games group: An active and passive behavior management will be applied by usage vid (Experimental)
  Interventions: Behavioral: Distraction

INTERVENTIONS:
Behavioral: Distraction — Control group: inferior alveolar nerve block will be administrated with passive behavior management (displaying animated movies directly on the screen of a mobile device).
  Movies group: inferior alveolar nerve block will be administrated with displaying animated movies directly on the screen of a mobile device usage of the augmented reality glasses.
  Video games group: Application of active behavior management by usage video games on the screen of a mobile device connected to augmented reality glasses before administration of inferior alveolar nerve block.
  Movies and Video games group: An active and passive behavior management will be applied by usage video games before administration of inferior alveolar nerve block and animated movies during administration on the screen of a mobile device connected to augmented reality glasses.

SUMMARY:
The aim of this study is to evaluate the effectiveness of augmented reality glasses in managing pain, anxiety, and behavior in pediatric patients during inferior alveolar nerve block

Group A (Control group): inferior alveolar nerve block will be administrated with passive behavior management (displaying animated movies directly on the screen of a mobile device).

Group B: inferior alveolar nerve block will be administrated with displaying animated movies directly on the screen of a mobile device usage of the augmented reality glasses.

Group C: Application of active behavior management by usage video games on the screen of a mobile device connected to augmented reality glasses before administration of inferior alveolar nerve block.

Group D: An active and passive behavior management will be applied by usage video games before administration of inferior alveolar nerve block and animated movies during administration on the screen of a mobile device connected to augmented reality glasses.

Children in all four groups will be assessed by using a combination of measures:

Venham's picture test (VPT), Pulse Oximeter, Wong-Baker face, observational behavioral scale (using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator") and general behavior scale (Houpt)

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of an augmented reality glasses. Pain, anxiety and general behavior will be evaluated during inferior alveolar nerve block using these behavioral scales, Venham's picture test (VPT), Pulse Oximeter, Wong-Baker face, observational behavioral scale (using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator") and general behavior scale (Houpt)

VPT scale consists of 8 associated drawings of a child, with each drawing showing a pair of children in two positions: non-anxious (value 0) and anxious (value 1). The child is asked to point to the child that expresses their feelings. The scale ranges from 0 to 8. If a child scores 6 or higher, they will be excluded from the research sample due to negative behavior. Anxiety is measured by monitoring pulse and oxygenation at five different times: before starting, 10 minutes later, when applying topical anesthetic, during the administration of the anesthetic injection, and immediately upon completion of the anesthetic injection. Using the Wong-Baker Faces scale to assess the level of pain after the anesthesia injection by asking the child to indicate the face that best represents their condition. The FLACC scale is a behavioral tool used to assess pain during the administration of an anesthesia injection. The child is recorded on video from before the injection starts until it is finished. The mobile phone is set up to film the child during the injection, and an external observer evaluates the child's behavior. The observer monitors five variables: (Face), (Legs), (Activity), (Cry), and (Consolability). Each variable is scored from 0 to 2, resulting in a total score ranging from 0 to 10. The Houpt scale was used to measure general behavior in children, as it consists of 6 points, starting from grade 1, which is the most violent behavior shown by the child during treatment, to grade 6, which is complete satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 7 and 9 years
2. Children categorized as having positive or definitely positive behavior on Frankl behavioral scale.
3. Children whose dental treatment requires an IANB injection.
4. Children with neither previous dental anesthesia experience nor augmented reality experience.
5. Children who do not suffer from any neurological, psychological or hearing disorders

Exclusion Criteria:

1. Children who refuse to put the glasses on.
2. Children suffering from acute dental pain.
3. Children suffering from auditory or visual disturbances

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Anxiety levels | before starting, ten minutes after stating, and after inferior alveolar nerve block injection
  VPT scale
Pain Levels | After administration of inferior alveolar nerve block
  Wong-Baker FACES
Pain Levels | after administration of topical anesthesia, during inferior alveolar nerve block injection, and directly after finishing of the injection]
  The Face-Legs-Activity-Cry-Consolability (FLACC) scale employing an external evaluator in which all of the body responses will be recorded during the administration of inferior alveolar nerve block. (0 low pain level - 10 highpain level)
Anxiety levels | before starting, ten minutes after stating, after administration of topical anesthesia, during inferior alveolar nerve block injection, and directly after finishing of the injection
  Pulse Oximeter

SECONDARY OUTCOMES:
General Behavior Level | during administration of inferior alveolar nerve block.
  Houpt scale consists of 6 points, starting from grade 1, which is the most violent behavior shown by the child during treatment, to grade 6, which is complete satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mai Maher Albaal, DDS, Principal Investigator — Department of Pediatric Dentistry, Faculty of Dentistry, University of Damascus, Damascus, Syria
Locations (1):
- Department of Pediatric Dentistry, Damascus, Syrian Arab Republic, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zafar S, Zachar JJ. Evaluation of HoloHuman augmented reality application as a novel educational tool in dentistry. Eur J Dent Educ. 2020 May;24(2):259-265. doi: 10.1111/eje.12492. Epub 2020 Jan 20. PMID 31899840
- [Background] Yeung AWK, Tosevska A, Klager E, Eibensteiner F, Laxar D, Stoyanov J, Glisic M, Zeiner S, Kulnik ST, Crutzen R, Kimberger O, Kletecka-Pulker M, Atanasov AG, Willschke H. Virtual and Augmented Reality Applications in Medicine: Analysis of the Scientific Literature. J Med Internet Res. 2021 Feb 10;23(2):e25499. doi: 10.2196/25499. PMID 33565986
- [Derived] Albaal M, Bshara N. Evaluating the use of augmented reality in alleviating anxiety and pain in children during intraoral injection administration: a randomized-controlled trial. Eur Arch Paediatr Dent. 2025 Sep 18. doi: 10.1007/s40368-025-01113-7. Online ahead of print. PMID 40965811